CLINICAL TRIAL: NCT06976788
Title: Creation of a Database of Healthy Subjects With 18FDG PET Brain Imaging as Part of the MOBILE Project (Multimodal Whole-Brain Imaging in Epilepsy)
Acronym: MOBILE-PET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RCAPHM22_0171
Record Dates: First submitted 2024-09-26; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-09

CONDITIONS: Healthy; Tomography; Brain Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole-Brain Imaging (Other)
  Interventions: Other: Tomography exam

INTERVENTIONS:
Other: Tomography exam — Brain imaging examination

SUMMARY:
The MOBILE project is part of the dynamic European collaboration of the Human Brain Project (HBP). The overall aim of the project is to characterize brain structure and function in healthy subjects and patients with epilepsy, using a quantitative multimodal approach involving both neuroimaging (MRI, PET) and electrophysiology (EEG/MEG). The project is funded by the European HBP consortium, and the data acquired will ultimately be made available to the scientific community formed by this international collaboration. Several aspects of the project have already been initiated on the basis of extensions to previous authorizations, or as part of care activities. As part of this overall project, the present MOBILE-PET application concerns exclusively the performance of 18F-FDG PET (Positron Emission Tomography) imaging in the 30 healthy adult subjects in the protocol (aged 18 to 65, with inclusion parity for gender). This cerebral examination, performed at rest on a 45-minute 3D volume acquisition, enables quantitative measurement of the metabolic consumption of glucose underlying global synaptic activity, and to determine the associated connectivity. Around 1,500 examinations of this type are carried out each year in our department as part of care for patients with brain pathology, and over 10,000 for patients with cancer. This examination requires intravenous injection of a weakly radioactive tracer corresponding to a radiopharmaceutical which has been approved for marketing for over 20 years. We also carried out and finalized a similar project in 2007 on 60 healthy subjects, using a previous-generation PET camera (NCT00484523). The Nuclear Medicine Department holds clinical research authorizations for imaging in patients and healthy subjects (including early phase and first-in-man, although the present project does not fall into this research categarogy).

ELIGIBILITY:
Inclusion Criteria:

* - Female or male, over 18 and under 65 years of age.
* Subject free of any general illness, psychiatric disorders or infectious, inflammatory, tumoral, vascular, degenerative or traumatic pathology of the central nervous system, as determined on examination,
* Subject not receiving chronic treatment, particularly psychotropic,
* Subject with no history of alcoholism or drug addiction,
* Subject with no contraindications to PET scintigraphic exploration (pregnancy and breast-feeding),
* Subject with social security coverage,
* Subject having read, understood and signed an informed consent form.

Exclusion Criteria:

* - Minors,
* Pregnant or breast-feeding women,
* Women of childbearing age without contraception,
* Subjects presenting a contraindication to PET scintigraphic exploration,
* adult subject to a legal protection measure, as provided for in L.1121-6 to L.1121-8 of the French Public Health Code.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
cerebral glucose consumption | Baseline and 24 months (longitudinal follow-up)

SECONDARY OUTCOMES:
Metabolic connectivity | Baseline and 24 months (longitudinal follow-up)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital de la Timone, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided